CLINICAL TRIAL: NCT04532060
Title: A Randomized Clinical Trial Evaluating Chlorine e6 Derivative-mediated Antimicrobial Photodynamic Therapy as a Treatment for Denture Stomatitis
Brief Title: Clinical Trial Evaluating Chlorine e6 Derivative-mediated Antimicrobial Photodynamic Therapy as a Treatment for Denture Stomatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: São Paulo State University (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FoAr
Record Dates: First submitted 2020-07-28; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Health Care Associated Infection
MeSH Terms: conditions — Cross Infection | interventions — Nystatin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antimicrobial Photodynamic Therapy (Experimental): Patients treated with Antimicrobial Photodynamic Therapy
  Interventions: Procedure: Antimicrobial Photodynamic Therapy
- Nystatin (Experimental): Patients treated with Nystatin antifungal drug.
  Interventions: Drug: Nystatin

INTERVENTIONS:
Drug: Nystatin
  Arms: Nystatin
Procedure: Antimicrobial Photodynamic Therapy
  Arms: Antimicrobial Photodynamic Therapy

SUMMARY:
Objective: This randomized clinical trial assessed antimicrobial Photodynamic Therapy (aPDT) mediated by Photodithazine (PDZ) to treat patients with denture stomatitis (DS). Methodologies: Patients with DS were randomly assigned to the groups: aPDT (n=30) and nystatin (NYS, n=35). aPDT patients received 6 aPDT sessions, three times a week for 15 days, which involved PDZ (200 mg/L) topical application (20 min) on the palate and upper denture, followed by light emitting diode (LED) illumination (660 nm, 50 J/cm²). NYS patients were instructed to rinse one dropper of this medication for one minute, four times a day, for 15 days. Microbiological collections of dentures and palates were performed and cultured on blood agar and CHROMAgar Candida. Microbial viability was determined, and photographs of the palates were taken for clinical evaluation. Data were analyzed by Repeated Measure Linear Model and Bonferroni (p≤0.05).

ELIGIBILITY:
Inclusion Criteria:

* Edentulous denture wearers clinically diagnosed with denture stomatitis.

Exclusion Criteria:

* patients who received antibiotics, antifungal or steroids in the past 3 months prior to the beginning of the research, women in the reproductive phase, patients who had worn the same denture in the past 10 years, diabetics, anemics, immunocompromised and under cancer treatment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2015-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Microbial Viability at baseline | The recovery of microorganisms was performed before the tretaments (at the baseline - initial).
  The efficacy of the treatments was verified microbiologically at the baseline (initial). For each patient, oral swabs were rubbed onto the palatal mucosa and on the tissue surface of the denture for 1 minute to recover the microorganisms. Each swab was placed into a Falcon tube (Corning, New York, USA) containing 5 mL of 0.9% sterile saline solution and vortexed for 1 minute to suspend the microorganisms from the swab. To evaluate Candida spp. survival and to presumptively identify Candida species by colony color, serial 10-fold dilutions from 100 to 103 were plated in duplicate on Chromagar Candida and incubated at 30 °C for 5 days. Additionally, to assess the total microbiota survival (fungal and bacteria), serial 10-fold dilutions from 102 to 104 were plated onto Blood agar.
Microbial Viability at the end of the treatments | The recovery of microorganisms was performed immediately at the end of the treatments.
  The efficacy of the treatments was verified microbiologically immediately at the end of the treatments. For each patient, oral swabs were rubbed onto the palatal mucosa and on the tissue surface of the denture for 1 minute to recover the microorganisms. Each swab was placed into a Falcon tube (Corning, New York, USA) containing 5 mL of 0.9% sterile saline solution and vortexed for 1 minute to suspend the microorganisms from the swab. To evaluate Candida spp. survival and to presumptively identify Candida species by colony color, serial 10-fold dilutions from 100 to 103 were plated in duplicate on Chromagar Candida and incubated at 30 °C for 5 days. Additionally, to assess the total microbiota survival (fungal and bacteria), serial 10-fold dilutions from 102 to 104 were plated onto Blood agar.
Microbial Viability on day 15 | The recovery of microorganisms was performed on day 15 after the end of the treatments.
  The efficacy of the treatments was verified microbiologically on day 15 after the end of the treatments. For each patient, oral swabs were rubbed onto the palatal mucosa and on the tissue surface of the denture for 1 minute to recover the microorganisms. Each swab was placed into a Falcon tube (Corning, New York, USA) containing 5 mL of 0.9% sterile saline solution and vortexed for 1 minute to suspend the microorganisms from the swab. To evaluate Candida spp. survival and to presumptively identify Candida species by colony color, serial 10-fold dilutions from 100 to 103 were plated in duplicate on Chromagar Candida and incubated at 30 °C for 5 days. Additionally, to assess the total microbiota survival (fungal and bacteria), serial 10-fold dilutions from 102 to 104 were plated onto Blood agar.
Microbial Viability on day 30 | The recovery of microorganisms was performed on day 30 after the end of the treatments.
  The efficacy of the treatments was verified microbiologically on day 30 after the end of the treatments. For each patient, oral swabs were rubbed onto the palatal mucosa and on the tissue surface of the denture for 1 minute to recover the microorganisms. Each swab was placed into a Falcon tube (Corning, New York, USA) containing 5 mL of 0.9% sterile saline solution and vortexed for 1 minute to suspend the microorganisms from the swab. To evaluate Candida spp. survival and to presumptively identify Candida species by colony color, serial 10-fold dilutions from 100 to 103 were plated in duplicate on Chromagar Candida and incubated at 30 °C for 5 days. Additionally, to assess the total microbiota survival (fungal and bacteria), serial 10-fold dilutions from 102 to 104 were plated onto Blood agar.
Microbial Viability on day 45 | The recovery of microorganisms was performed on day 45 after the end of the treatments.
  The efficacy of the treatments was verified microbiologically on day 45 after the end of the treatments. For each patient, oral swabs were rubbed onto the palatal mucosa and on the tissue surface of the denture for 1 minute to recover the microorganisms. Each swab was placed into a Falcon tube (Corning, New York, USA) containing 5 mL of 0.9% sterile saline solution and vortexed for 1 minute to suspend the microorganisms from the swab. To evaluate Candida spp. survival and to presumptively identify Candida species by colony color, serial 10-fold dilutions from 100 to 103 were plated in duplicate on Chromagar Candida and incubated at 30 °C for 5 days. Additionally, to assess the total microbiota survival (fungal and bacteria), serial 10-fold dilutions from 102 to 104 were plated onto Blood agar.

SECONDARY OUTCOMES:
Clinical evaluation | Standardized photographs of the palates were taken prior to the beginning of the treatments (initial) and up to 45 days after the end of the treatments.
  To verify the clinical efficacy of the treatments, the oral lesions on the palatal mucosal were evaluated. For this, standardized photographs of the palates were taken prior to the beginning of the treatments (initial) and up to 45 days after the end of the treatments. All the photographs were taken with the same digital camera (NIKON D7000, Tokyo, Japan), by the same operator, under the same conditions (place, light, position). After that, all photographs were analyzed by two individuals blinded to the treatment performed, to classify the oral lesion in type I, II or III in all time intervals.

IPD SHARING:
Plan to Share IPD: No